CLINICAL TRIAL: NCT06944470
Title: JS207 (Anti-PD-1/VEGF Bispecific Antibody) Combined With Platinum-based Doublet Chemotherapy in Subjects With Stage II-III Non-small Cell Lung Cancer
Brief Title: JS207 Combined With Chemotherapy in Subjects With Stage II-III NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS207-005-II-NSCLC
Record Dates: First submitted 2025-04-15; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: NSCLC
MeSH Terms: interventions — Paclitaxel; Carboplatin; Cisplatin; Pemetrexed; Surgical Procedures, Operative; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort1：enrolled untreated resectable stage II-III NSCLC patients（JS207） (Experimental): Preoperative neoadjuvant therapy phase, the receive JS207 + platinum-based double chemotherapyonce every 3 weeks，then perform Surgical treatment，after that，perform postoperative ADJUVANT THERAPY （JS207）
  Interventions: Drug: Paclitaxel + Carboplatin/cisplatin for squamous cell carcinoma and pemetrexed + carboplatin/cisplatin for non-squamous cell carcinoma; Procedure: surgery; Drug: JS207
- Cohort2：enrolled untreated, stage III NSCLC patients（JS207） (Experimental): Preoperative neoadjuvant therapy phase, the receive JS207 + platinum-based double chemotherapyonce every 3 weeks，then perform Surgical treatment or CRT，after that，perform postoperative ADJUVANT THERAPY （JS207）
  Interventions: Drug: Paclitaxel + Carboplatin/cisplatin for squamous cell carcinoma and pemetrexed + carboplatin/cisplatin for non-squamous cell carcinoma; Procedure: surgery; Radiation: Radiochemotherapy; Drug: JS207

INTERVENTIONS:
Drug: Paclitaxel + Carboplatin/cisplatin for squamous cell carcinoma and pemetrexed + carboplatin/cisplatin for non-squamous cell carcinoma — Carboplatin Injection:
  One dose of carboplatin AUC 5 IV on Day 1 of each 3-week cycle.
  Cisplatin injection:
  Cisplatin 75 mg/m2 IV on Day 1 of every 3-week cycle.
  Paclitaxel injection:
  175 mg/m2 IV on Day 1 of each 3-week cycle.
  Pemetrexed Injection:
  Pemetrexed 500 mg/m2 IV on Day 1 of each 3-week cycle.
Procedure: surgery — Subjects with surgical indications will undergo radical surgery for NSCLC，within 4-6 weeks after the last dose of neoadjuvant therapy.
Radiation: Radiochemotherapy — If radical surgery is not suitable after MDT evaluation, the subjects will receive comprehensive treatment mainly based on radiotherapy.
  Arms: Cohort2：enrolled untreated, stage III NSCLC patients（JS207）
Drug: JS207 — JS207 will be administered every 3 weeks for a treatment cycle of 21 days.

SUMMARY:
This is a phase II clinical study to evaluate the safety, tolerability, preliminary efficacy and pharmacokinetics of JS207 (anti-PD-1/VEGF bispecific antibody) combined with platinum-based doublet chemotherapy in subjects with stage II-III non-small cell lung cancer. The study consists of 2 cohorts, including treatment-naïve and resectable subjects with stage II-III NSCLC (cohort 1), treatment-naïve and unresectalbe subjects with stage III NSCLC (cohort 2). Subjects in both cohorts will receive 3 cycles of JS207 + platinum-based doublet chemotherapy as neoadjuvant therapy, followed by surgery or definitive chemoradiotherapy, and then adjuvant therapy with JS207 (post-surgery) or consolidation therapy with JS207 (post-chemoradiotherapy).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years at the time of signing the informed consent (inclusive of 18 and 75 years), either gender.
2. Histologically confirmed, previously untreated stage II-III NSCLC (AJCC 8th edition), cTNM stage can be confirmed by PET-CT or pathological biopsy. For suspicious lesions that are suspected by imaging examination, which can lead to changes in TNM stage, including but not limited to contralateral mediastinal lymph nodes and supraclavicular lymph nodes, pathological biopsy verification is strongly recommended.

   1. Cohort 1: Subjects with resectable, stage II, IIIA, or IIIB (N2) NSCLC evaluated by MDT.
   2. Cohort 2: Subjects with unresectable, stage III NSCLC evaluated by MDT.
3. Total lung function can withstand the proposed lung resection procedure according to the surgeon's evaluation.
4. Subjects without EGFR sensitive mutation, ALK fusion, ROS1 fusion or RET fusion. Subjects with squamous cell carcinoma are not required to undergo genetic testing. The Certificate of Analysis from the local laboratory is acceptable, but the test must be well validated and approved by the inter-laboratory quality assessment or NMPA (if the mutation is negative in blood test, it must be confirmed based on the results from tissue sample); if there is no previous Certificate of Analysis or the previous Certificate of Analysis does not meet the requirements, the sample should be provided for testing.
5. At least 3 unstained tumor tissue sections were available for detection of PD-L1 and other biomarkers. If truly unable to provide tumor tissue samples as required, enrollment was also possible after communication with the sponsor.
6. Function of vital organs meets the requirements.

Exclusion Criteria:

1. In the company of the following study disease status:

   1. Histopathologically or cytologically confirmed combined components of neuroendocrine tumours (including small cell lung cancer, large cell neuroendocrine carcinoma, etc.) and Pancoast tumor.
   2. Tumor encircles important blood vessels or has obvious necrosis and air space, and the investigator considers that it may cause hemorrhage risk.
   3. Any clinically significant hemoptysis (≥2.5 ml) or Tumour haemorrhage of any cause within one month before the first use of the study drug.
2. Received any of the following treatments:

   1. Previous systemic antitumor therapy for NSCLC (including investigational drugs), such as chemotherapy or immunologically mediated therapy (including but not limited to anti-PD-1, anti-PD-L1, anti-CTLA-4 therapy) and anti-angiogenic therapy (such as anti-VEGF pathway-targeted drugs);
   2. Prior radiotherapy to chest;
3. History of significant Haemorrhagic diathesis or severe Disorder coagulation, or Grade ≥3 bleeding event within 6 months prior to the first dose, or current ≥Grade 2 bleeding or factors that are judged by the investigator to be at high risk for bleeding (e.g., active peptic ulcer or Varices oesophageal).
4. Gastrointestinal perforation, intra-abdominal fistula, or intra-abdominal abscess within 6 months prior to the first dose, or current risk factors for perforation/fistula formation of hollow organs as judged by the investigator, such as tumor invasion of the outer layer of hollow organ wall, or active inflammatory bowel disease (including Colitis ulcerative and Crohn's disease), Diverticulitis, Cholecystitis, symptomatic Cholangitis or Appendicitis.
5. Existence of poorly controlled Hypertension, or history of Hypertensive crisis or Hypertensive encephalopathy.
6. Active autoimmune disease, history of autoimmune disease (such as interstitial pneumonitis, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); except Vitiligo or childhood asthma/allergy that has been cured, patients who do not require any intervention after adulthood, patients with autoimmune-mediated hypothyroidism treated with a stable dose of thyroid replacement hormone, patients with hyperthyroidism adequately treated and well-controlled, and patients with type I Diabetes mellitus treated with a stable dose of Insulin, etc.
7. Uncontrolled co-morbidities, including but not limited to: symptomatic congestive heart failure, left ventricular ejection fraction (LVEF) <50%, unstable angina, treated arrhythmia, aortic aneurysm requiring surgical repair, any arterial thrombotic/embolic events, Grade 3 or higher (CTCAE 5.0) venous thrombotic/embolic events, transient ischemic attack, cerebrovascular accident, tracheoesophageal fistula, gastrointestinal perforation, intra-abdominal abscess, gastrointestinal obstruction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
PCR rate | 2 years
  To evaluate the pathologic complete response rate (pCR rate) of JS207 combined with platinum-based doublet chemotherapy in subjects with resectable stage II-III NSCLC and subjects with uresectable stage III NSCLC.

SECONDARY OUTCOMES:
MPR rate | 2 years
  To evaluate the pathologic MPR rate of JS207 combined with platinum-based doublet chemotherapy in subjects with resectable stage II-III NSCLC and subjects with uresectable stage III NSCLC.
EFS | 2 years
  Time from the beginning of randomization until disease progression under the RECIST1.1 criteria is first recorded leading to inoperable or CRT, local progression leading to inoperable tumor resection or CRT, CRT or postoperative disease recurrence or progression, or death from any cause, whichever occurs first
ORR | 2 years
  Subjects with partial response (PR) or complete response (CR) at BOR
DCR | 2 years
  Proportion of subjects with CR, PR, or stable disease (SD) at BOR
OS | 2 years
  The time from first dose to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No